CLINICAL TRIAL: NCT04019990
Title: The Effect of Thrower's Ten Exercise Programme On Upper Extremity Muscle Power, Range of Motion and Explosive Power in Wheelchair Basketball and Basketball Players
Brief Title: Throwers Ten Exercises On Upper Extremity Function and Explosive Power in Wheelchair Basketball and Basketball Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ceyda Sofuoğlu, Principal investigator, Hacettepe University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: GO15/204
Record Dates: First submitted 2019-07-07; First posted 2019-07-15 (Actual); Results first posted 2020-02-12 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-02

CONDITIONS: Upper Extremity Injury; Sport Injury; Shoulder Pain; Muscle Weakness
Keywords: Sports for Persons with Disabilities; Basketball; Exercise
MeSH Terms: conditions — Arm Injuries; Shoulder Pain; Muscle Weakness; Motor Activity

STUDY DESIGN:
Intervention Model Description: 13 players from the North Cyprus wheelchair Basketball Team and 15 players from the Koop Bank Basketball Men's Team voluntarily will participate in the study. Subjects will include to study if they fulfil criteria. J-Tech medical tracker freedom will use for measuring upper extremity muscle power and range of motion. Medicine ball throw test will use for plyometric power. Athletes will involve in 8 weeks Thrower's Ten exercise program. After 8. Weeks and 12. Weeks assessments will be repeated.
  The exercise programme will conduct 3 days a week, with 2 days a week as a group under the supervision of a physiotherapist in the rehabilitation center and 1 day at the homes of the participants without any supervision. The home programme will be monitored by contacting the players over the telephone. The training is planned to progress every 3 weeks, and progression programme will plan individually according to player progression.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Wheelchair basketball and ambulant basketball players (Other): 13 players from the North Cyprus wheelchair Basketball Team and 15 players from the Koop Bank Basketball Men's Team voluntarily will participate in the study. Subjects will include to study if they fulfil criteria. Athletes will involve in 8 weeks Thrower's Ten exercise program. After 8. Weeks and 12. Weeks assessments will be repeated.
  Interventions: Other: The effect of throwers ten exercise programme on wheelchair basketball and ambulant basketball players

INTERVENTIONS:
Other: The effect of throwers ten exercise programme on wheelchair basketball and ambulant basketball players — Throwers Ten exercise programme is a programme designed to improve the power, strength and endurance of large muscle groups required for the throwing activity. It consists of exercises involving the movement of upper limb joints in full range of joint motion or at specified specific angles, with the help of a resistance band and weights specific to individual athletes. In the literature, no study has demonstrated the effectiveness of Throwers Ten exercise programme in wheelchair basketball and ambulant basketball players.

SUMMARY:
Basketball is a challenging sport that requires participants to demonstrate physical fitness and special athletic skills at high levels. Players avoid contact while attempting to prevent the opponent from running, passing and shooting. Although basketball includes avoiding contact as a rule, contact between players is inevitable. Various injuries occur in basketball because it is a contact sport and includes sudden movements, such as bouncing, running and turning. Wheelchair (WC) basketball is characterised by manoeuvres and high-intensity activities such as rolling, rebounding, passing and overhead shooting. In WC basketball players, thoracic kyphosis is increased because of atrophy of the upper back and shoulders muscles resulting from the body posture required for WC propulsion in the sitting position as well as the effect of gravity. This sitting posture is characterised by scapular protraction and internal rotation of the humerus, and it impedes shoulder movements during upper-extremity use.

Overhead throwing is a movement that involves high speed and repetitive movement that leads to upper-extremity injuries. It is important to develop muscle strength and proprioception to protect against these injuries.

Throwers Ten exercise programme is a programme designed to improve the power, strength and endurance of large muscle groups required for the throwing activity. It consists of exercises involving the movement of upper limb joints in full range of joint motion (ROM) or at specified specific angles, with the help of a resistance band and weights specific to individual athletes.

In the literature, no study has demonstrated the effectiveness of Throwers Ten exercise programme in these sports groups. The aim of this study was to evaluate the effectiveness of Throwers Ten exercise programme on upper-extremity function and explosive power in the WC basketball players and stand-up basketball players.

DETAILED DESCRIPTION:
Basketball is a challenging sport that requires participants to demonstrate physical fitness and special athletic skills at high levels. Players avoid contact while attempting to prevent the opponent from running, passing and shooting. Although basketball includes avoiding contact as a rule, contact between players is inevitable. Various injuries occur in basketball because it is a contact sport and includes sudden movements, such as bouncing, running and turning.

Wheelchair (WC) basketball is characterised by manoeuvres and high-intensity activities such as rolling, rebounding, passing and overhead shooting. In WC basketball players, thoracic kyphosis is increased because of atrophy of the upper back and shoulders muscles resulting from the body posture required for WC propulsion in the sitting position as well as the effect of gravity. This sitting posture is characterised by scapular protraction and internal rotation of the humerus, and it impedes shoulder movements during upper-extremity use. The force balance changes because of humeral internal rotation and scapular protraction, and the internal rotator and adductor muscles become stronger than their antagonists. In basketball, throwing and pushing are used to pass the ball to the target. In throwing, the force of the dominant upper extremity comes into play with the internal rotation of the humerus. In this movement, the humerus is almost horizontal and parallel to the ground.

Increased use of the upper extremities in WC users increases upper-extremity load. For this reason, upper-extremity muscle strength, endurance and explosive power are of great importance. Rotational muscle strength of the shoulder has critical roles in activities specific to basketball as well as WC control in WC basketball players.

Overhead throwing is a movement that involves high speed and repetitive movement that leads to upper-extremity injuries. It is important to develop muscle strength and proprioception to protect against these injuries.

Throwers Ten exercise programme is a programme designed to improve the power, strength and endurance of large muscle groups required for the throwing activity. It consists of exercises involving the movement of upper limb joints in full range of joint motion (ROM) or at specified specific angles, with the help of a resistance band and weights specific to individual athletes. In a study conducted by Wilk et al., it was reported that muscle strength and endurance were improved by increasing muscle activation and facilitation, and achieving dynamic stabilisation by adding isometric contractions to the concentric/eccentric contractions applied in the Throwers Ten exercise programme.

In the literature, no study has demonstrated the effectiveness of Throwers Ten exercise programme in these sports groups. The aim of this study was to evaluate the effectiveness of Throwers Ten exercise programme on upper-extremity function and explosive power in the WC basketball players and stand-up basketball players. In addition, because the WC basketball players and stand-up basketball players were evaluated in this study, our secondary aim was to elucidate the differences in responses to the exercise programme between a group without lower-extremity use and incomplete strength distribution and a group with complete strength distribution.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic athletes
* Professional athlete who plays at least 10 years
* Subjects who are voluntary to participate in the study

Exclusion Criteria:

* Upper extremity related surgery in past 6 months
* Rotator cuff tears in past 3 months
* Current pain in shoulder and neck

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-11-20 (Actual); Study Completion 2019-11-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Volga Bayrakcı Tunay, Study Director — Hacettepe University
Locations (1):
- Mehmet Reis Physiotherapy and Rehabilitation Center, Nicosia, Lefkoşa, Cyprus

IPD SHARING:
Plan to Share IPD: Yes
IPD data for all primary and secondary measures will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available within 1 year of study completion.
Access Criteria: Data access requests will be reviewed by an external İndependent Review Panel. Requestors will be required to sign a Data Access Agreement.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: During evaluations and training, 1 wheelchair basketball player, and 3 stand-up basketball players were excluded from the study as they failed to meet the inclusion criteria.
Groups:
- Wheelchair Basketball Players: 13 players from the North Cyprus Turkcell Wheelchair Basketball Team voluntarily participated in the study. During evaluations and training, one WC basketball player was excluded from the study as they failed to meet the inclusion criteria. After preliminary evaluation, all participants took part in the Throwers Ten exercise programme 3 days a week for 8 weeks. Evaluations were made before the exercise programme, at week 8 at programme completion, and at week 12 after programme completion.
- Ambulant Basketball Players: 15 players from the Koop Bank Basketball Men's Team voluntarily participated in the study. During evaluations and training three basketball players were excluded from the study as they failed to meet the inclusion criteria. After preliminary evaluation, all participants took part in the Throwers Ten exercise programme 3 days a week for 8 weeks. Evaluations were made before the exercise programme, at week 8 at programme completion, and at week 12 after programme completion.
Period: Overall Study
Arm/Group | Wheelchair Basketball Players | Ambulant Basketball Players
Started | 13 | 15
Completed | 12 | 12
Not Completed | 1 | 3

BASELINE CHARACTERISTICS:
Population: During evaluations and training, 1 WC basketball player, and 3 stand-up basketball players were excluded from the study as they failed to meet the inclusion criteria.
Arm/Group | Wheelchair Basketball and Ambulant Basketball Players
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 22
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 24
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Cypriot | 24
Region of Enrollment [Count of Participants; unit: Participants]
  Cyprus | 24
Sporting Experience (year) [Mean (Standard Deviation); unit: years] — Population: 12 Wheelchair Basketball players and 12 Ambulant Basketball players were analyzed. Because of that there are 2 row population and the overall number is 24.
  years
    Wheelchair Basketball Players: number analyzed (Participants) | 12
    Wheelchair Basketball Players | 10.6 (6.9)
    Ambulant Basketball Players: number analyzed (Participants) | 12
    Ambulant Basketball Players | 12.2 (8.1)
Body Mass İndex (kg/m²) [Mean (Standard Deviation); unit: kg/m²] — Population: 12 Wheelchair Basketball players and 12 Ambulant Basketball players were analyzed. Because of that there are 2 row population and the overall number is 24.
  kg/m²
    Wheelchair Basketball Players: number analyzed (Participants) | 12
    Wheelchair Basketball Players | 23.18 (4.63)
    Ambulant Basketball Players: number analyzed (Participants) | 12
    Ambulant Basketball Players | 25.46 (0.9)

OUTCOME MEASURES:

1. Primary Outcome: Measurement of Muscle Strength (Absolute Values Are Being Reported)
Description: The strength of shoulder flexion, abduction, external rotation (E.R), internal rotation(İ.R) and elbow flexion will measure as isometric muscle strength in kg by J-Tech Medical/USA Tracker Freedom Isometric Muscle Test.
Time Frame: All measurements will repeat three times at 5-s intervals and the mean value will be taken. Baseline, 8 and 12 Weeks reported.
Population: 12 Wheelchair basketball players and 12 ambulant basketball players muscle strength test results in baseline, 8 Week and 12 Week were compared.
Measure: Mean (Standard Deviation); unit: kg
Groups:
- Wheelchair Basketball and Ambulant Basketball Players: 13 players from the North Cyprus Turkcell Wheelchair Basketball Team and 15 players from the Koop Bank Basketball Men's Team voluntarily participated in the study. During evaluations and training, 1 wheelchair basketball player, and 3 stand-up basketball players were excluded from the study as they failed to meet the inclusion criteria. The final participants were 12 male wheelchair basketball players and12 male stand-up basketball players. After preliminary evaluation, all participants took part in the Throwers Ten exercise programme 3 days a week for 8 weeks. Evaluations were made before the exercise programme, at week 8 at programme completion, and at week 12 after programme completion.
Arm/Group | Wheelchair Basketball and Ambulant Basketball Players
Number analyzed (Participants) | 24
kg
  ShoulderFlexionWheelchairBasketballRight Baseline: number analyzed (Participants) | 12
  ShoulderFlexionWheelchairBasketballRight Baseline | 3.9 (0.7)
  ShoulderFlexionAmbulantBasketballRight Baseline: number analyzed (Participants) | 12
  ShoulderFlexionAmbulantBasketballRight Baseline | 5.1 (0.9)
  ShoulderFlexionWheelchairBasketballRight at 8 Week: number analyzed (Participants) | 12
  ShoulderFlexionWheelchairBasketballRight at 8 Week | 5.7 (1.5)
  ShoulderFlexionAmbulantBasketballRight at 8 Week: number analyzed (Participants) | 12
  ShoulderFlexionAmbulantBasketballRight at 8 Week | 7.4 (1.5)
  ShoulderFlexionWheelchairBasketballRight at 12Week: number analyzed (Participants) | 12
  ShoulderFlexionWheelchairBasketballRight at 12Week | 5.5 (1.6)
  ShoulderFlexionAmbulantBasketballRight at 12 Week: number analyzed (Participants) | 12
  ShoulderFlexionAmbulantBasketballRight at 12 Week | 5.4 (0.8)
  ShoulderFlexionWheelchairBasketball Left Baseline: number analyzed (Participants) | 12
  ShoulderFlexionWheelchairBasketball Left Baseline | 3.8 (0.7)
  ShoulderFlexionAmbulantBasketball Left at Baseline: number analyzed (Participants) | 12
  ShoulderFlexionAmbulantBasketball Left at Baseline | 5.5 (0.8)
  ShoulderFlexionWheelchairBasketball Left at 8 Week: number analyzed (Participants) | 12
  ShoulderFlexionWheelchairBasketball Left at 8 Week | 5.7 (1.8)
  ShoulderFlexionAmbulantBasketball Left at 8 Week: number analyzed (Participants) | 12
  ShoulderFlexionAmbulantBasketball Left at 8 Week | 7.5 (1)
  ShoulderFlexionWheelchairBasketball Left at 12Week: number analyzed (Participants) | 12
  ShoulderFlexionWheelchairBasketball Left at 12Week | 5.5 (1.8)
  ShoulderFlexionAmbulantBasketball Left at 12 Week: number analyzed (Participants) | 12
  ShoulderFlexionAmbulantBasketball Left at 12 Week | 5.8 (0.8)
  ShoulderAbductionWheelchairBasketballRightBaseline: number analyzed (Participants) | 12
  ShoulderAbductionWheelchairBasketballRightBaseline | 4 (0.7)
  ShoulderAbductionAmbulantBasketballRight Baseline: number analyzed (Participants) | 12
  ShoulderAbductionAmbulantBasketballRight Baseline | 5.4 (1.2)
  ShoulderAbductionWheelchairBasketballRight at8Week: number analyzed (Participants) | 12
  ShoulderAbductionWheelchairBasketballRight at8Week | 5.9 (1.7)
  ShoulderAbductionAmbulantBasketballRight at8Week: number analyzed (Participants) | 12
  ShoulderAbductionAmbulantBasketballRight at8Week | 7.4 (1.3)
  ShoulderAbductionWheelchairBasketballRightat12Week: number analyzed (Participants) | 12
  ShoulderAbductionWheelchairBasketballRightat12Week | 5.7 (1.7)
  ShoulderAbductionAmbulantBasketballRight at12Week: number analyzed (Participants) | 12
  ShoulderAbductionAmbulantBasketballRight at12Week | 5.8 (1.2)
  ShoulderAbductionWheelcahairBasketballLeftBaseline: number analyzed (Participants) | 12
  ShoulderAbductionWheelcahairBasketballLeftBaseline | 3.7 (0.7)
  ShoulderAbductionAmbulantBasketballLeft Baseline: number analyzed (Participants) | 12
  ShoulderAbductionAmbulantBasketballLeft Baseline | 5.8 (0.8)
  ShoulderAbductionWheelchairBasketballLeft at8Week: number analyzed (Participants) | 12
  ShoulderAbductionWheelchairBasketballLeft at8Week | 5.9 (1.7)
  ShoulderAbductionAmbulantBasketballLeft at8Week: number analyzed (Participants) | 12
  ShoulderAbductionAmbulantBasketballLeft at8Week | 7.7 (1)
  ShoulderAbductionWheelchairBasketballLeft at12Week: number analyzed (Participants) | 12
  ShoulderAbductionWheelchairBasketballLeft at12Week | 5.7 (1.7)
  ShoulderAbductionAmbulantBasketballLeft at12Week: number analyzed (Participants) | 12
  ShoulderAbductionAmbulantBasketballLeft at12Week | 6.2 (1)
  Shoulder E.R WheelchairBasketball Right Baseline: number analyzed (Participants) | 12
  Shoulder E.R WheelchairBasketball Right Baseline | 1.8 (0.4)
  Shoulder E.R Ambulant Basketball Right Baseline: number analyzed (Participants) | 12
  Shoulder E.R Ambulant Basketball Right Baseline | 3.9 (0.8)
  Shoulder E.R WheelchairBasketball Right at 8 Week: number analyzed (Participants) | 12
  Shoulder E.R WheelchairBasketball Right at 8 Week | 4.4 (1.6)
  Shoulder E.R Ambulant Basketball Right at 8 Week: number analyzed (Participants) | 12
  Shoulder E.R Ambulant Basketball Right at 8 Week | 4.9 (1.1)
  Shoulder E.R WheelchairBasketball Right at 12 Week: number analyzed (Participants) | 12
  Shoulder E.R WheelchairBasketball Right at 12 Week | 4.1 (1.6)
  Shoulder E.R Ambulant Basketball Right at 12 Week: number analyzed (Participants) | 12
  Shoulder E.R Ambulant Basketball Right at 12 Week | 4.2 (0.7)
  Shoulder E.R WheelchairBasketball Left Baseline: number analyzed (Participants) | 12
  Shoulder E.R WheelchairBasketball Left Baseline | 1.8 (0.4)
  Shoulder E.R Ambulant Basketball Left Baseline: number analyzed (Participants) | 12
  Shoulder E.R Ambulant Basketball Left Baseline | 4.1 (0.6)
  Shoulder E.R WheelchairBasketball Left at 8 Week: number analyzed (Participants) | 12
  Shoulder E.R WheelchairBasketball Left at 8 Week | 4.5 (1.7)
  Shoulder E.R Ambulant Basketball Left at 8 Week: number analyzed (Participants) | 12
  Shoulder E.R Ambulant Basketball Left at 8 Week | 4.9 (0.9)
  Shoulder E.R WheelchairBasketball Left at 12 Week: number analyzed (Participants) | 12
  Shoulder E.R WheelchairBasketball Left at 12 Week | 4.3 (1.6)
  Shoulder E.R Ambulant Basketball Left at 12 Week: number analyzed (Participants) | 12
  Shoulder E.R Ambulant Basketball Left at 12 Week | 4.5 (0.7)
  Shoulder İ.R WheelchairBasketball Right Baseline: number analyzed (Participants) | 12
  Shoulder İ.R WheelchairBasketball Right Baseline | 1.9 (0.4)
  Shoulder İ.R Ambulant Basketball Right Baseline: number analyzed (Participants) | 12
  Shoulder İ.R Ambulant Basketball Right Baseline | 4.8 (1)
  Shoulder İ.R WheelchairBasketball Right at 8 Week: number analyzed (Participants) | 12
  Shoulder İ.R WheelchairBasketball Right at 8 Week | 5.5 (2.3)
  Shoulder İ.R Ambulant Basketball Right at 8 Week: number analyzed (Participants) | 12
  Shoulder İ.R Ambulant Basketball Right at 8 Week | 6.6 (1)
  Shoulder İ.R WheelchairBasketball Right at 12 Week: number analyzed (Participants) | 12
  Shoulder İ.R WheelchairBasketball Right at 12 Week | 5.3 (2.4)
  Shoulder İ.R Ambulant Basketball Right at 12 Week: number analyzed (Participants) | 12
  Shoulder İ.R Ambulant Basketball Right at 12 Week | 5.3 (1.3)
  Shoulder İ.R WheelchairBasketball Left Baseline: number analyzed (Participants) | 12
  Shoulder İ.R WheelchairBasketball Left Baseline | 1.9 (0.5)
  Shoulder İ.R Ambulant Basketball Left Baseline: number analyzed (Participants) | 12
  Shoulder İ.R Ambulant Basketball Left Baseline | 3.8 (0.7)
  Shoulder İ.R WheelchairBasketball Left at 8 Week: number analyzed (Participants) | 12
  Shoulder İ.R WheelchairBasketball Left at 8 Week | 4.4 (1.7)
  Shoulder İ.R Ambulant Basketball Left at 8 Week: number analyzed (Participants) | 12
  Shoulder İ.R Ambulant Basketball Left at 8 Week | 5.5 (0.8)
  Shoulder İ.R WheelchairBasketball Left at 12 Week: number analyzed (Participants) | 12
  Shoulder İ.R WheelchairBasketball Left at 12 Week | 4.2 (1.7)
  Shoulder İ.R Ambulant Basketball Left at 12 Week: number analyzed (Participants) | 12
  Shoulder İ.R Ambulant Basketball Left at 12 Week | 4.1 (0.9)
  Elbow Flexion WheelchairBasketball Right Baseline: number analyzed (Participants) | 12
  Elbow Flexion WheelchairBasketball Right Baseline | 3 (0.8)
  Elbow Flexion Ambulant Basketball Right Baseline: number analyzed (Participants) | 12
  Elbow Flexion Ambulant Basketball Right Baseline | 6.6 (1.1)
  Elbow Flexion WheelchairBasketball Right at 8 Week: number analyzed (Participants) | 12
  Elbow Flexion WheelchairBasketball Right at 8 Week | 6.7 (2.6)
  Elbow Flexion Ambulant Basketball Right at 8 Week: number analyzed (Participants) | 12
  Elbow Flexion Ambulant Basketball Right at 8 Week | 7.7 (1.1)
  Elbow Flexion WheelchairBasketball Right at 12Week: number analyzed (Participants) | 12
  Elbow Flexion WheelchairBasketball Right at 12Week | 6.2 (2.3)
  Elbow Flexion Ambulant Basketball Right at 12 Week: number analyzed (Participants) | 12
  Elbow Flexion Ambulant Basketball Right at 12 Week | 6.9 (1.3)
  Elbow Flexion WheelchairBasketball Left Baseline: number analyzed (Participants) | 12
  Elbow Flexion WheelchairBasketball Left Baseline | 2.6 (0.5)
  Elbow Flexion Ambulant Basketball Left Baseline: number analyzed (Participants) | 12
  Elbow Flexion Ambulant Basketball Left Baseline | 6.3 (0.8)
  Elbow Flexion WheelchairBasketball Left at 8 Week: number analyzed (Participants) | 12
  Elbow Flexion WheelchairBasketball Left at 8 Week | 6 (2.7)
  Elbow Flexion Ambulant Basketball Left at 8 Week: number analyzed (Participants) | 12
  Elbow Flexion Ambulant Basketball Left at 8 Week | 7.5 (1.2)
  Elbow Flexion WheelchairBasketball Left at 12 Week: number analyzed (Participants) | 12
  Elbow Flexion WheelchairBasketball Left at 12 Week | 5.7 (2.7)
  Elbow Flexion Ambulant Basketball Left at 12 Week: number analyzed (Participants) | 12
  Elbow Flexion Ambulant Basketball Left at 12 Week | 6.5 (0.7)

2. Primary Outcome: Medicine Ball Throwing Test (Absolute Values Are Being Reported)
Description: In this test, the distance that a 3-kg ball can be thrown will measure to assess upper-extremity explosive strength. The test will conduct in two different positions. In the first test, the participant will seat in a chair of sufficient height without armrests so that the scapula will be in a free position. The ball is then grasp with both hands and throw forward overhead, and the distance will record. In the second test, the participant is in the same starting position and throw the ball forward with two hands after bringing it to the chest level, and the distance will record.
Time Frame: as for outcome 1
Population: 12 Wheelchair basketball (W.B) players and 12 ambulant basketball (A.B) players medicine ball throwing test results in Baseline, 8 Weeks and 12 Weeks were compared.
Measure: Mean (Standard Deviation); unit: cm
Groups:
- Wheelchair Basketball and Ambulant Basketball Players: 13 players from the North Cyprus Turkcell Wheelchair Basketball Team and 15 players from the Koop Bank Basketball Men's Team voluntarily participated in the study. During evaluations and training, one WC basketball player, and three stand-up basketball players were excluded from the study as they failed to meet the inclusion criteria. The final participants were 12 male wheelchair basketball players and 12 male stand-up basketball players. After preliminary evaluation, all participants took part in the Throwers Ten exercise programme 3 days a week for 8 weeks. Evaluations were made before the exercise programme, at week 8 at programme completion, and at week 12 after programme completion.
Arm/Group | Wheelchair Basketball and Ambulant Basketball Players
Number analyzed (Participants) | 24
cm
  Medicine Ball Overhead Throw W.B Baseline: number analyzed (Participants) | 12
  Medicine Ball Overhead Throw W.B Baseline | 360.6 (103.8)
  Medicine Ball Overhead Throw A.B Baseline: number analyzed (Participants) | 12
  Medicine Ball Overhead Throw A.B Baseline | 603.5 (73.4)
  Medicine Ball Overhead Throw W.B 8 Week: number analyzed (Participants) | 12
  Medicine Ball Overhead Throw W.B 8 Week | 386.9 (110.1)
  Medicine Ball Overhead Throw A.B 8 Week: number analyzed (Participants) | 12
  Medicine Ball Overhead Throw A.B 8 Week | 606.2 (100.5)
  Medicine Ball Overhead Throw W.B 12 Week: number analyzed (Participants) | 12
  Medicine Ball Overhead Throw W.B 12 Week | 370 (104.6)
  Medicine Ball Overhead Throw A.B 12 Week: number analyzed (Participants) | 12
  Medicine Ball Overhead Throw A.B 12 Week | 599.3 (82.1)
  Medicine Ball Chest Throw W.B Baseline: number analyzed (Participants) | 12
  Medicine Ball Chest Throw W.B Baseline | 410.3 (142)
  Medicine Ball Chest Throw A.B Baseline: number analyzed (Participants) | 12
  Medicine Ball Chest Throw A.B Baseline | 597.2 (64.4)
  Medicine Ball Chest Throw W.B 8 Week: number analyzed (Participants) | 12
  Medicine Ball Chest Throw W.B 8 Week | 439.4 (147.6)
  Medicine Ball Chest Throw A.B 8 Week: number analyzed (Participants) | 12
  Medicine Ball Chest Throw A.B 8 Week | 645.8 (50.6)
  Medicine Ball Chest Throw W.B 12 Week: number analyzed (Participants) | 12
  Medicine Ball Chest Throw W.B 12 Week | 421.5 (146.7)
  Medicine Ball Chest Throw A.B 12 Week: number analyzed (Participants) | 12
  Medicine Ball Chest Throw A.B 12 Week | 605.7 (60)

3. Primary Outcome: Hand Grip Test (Absolute Value Are Being Reported)
Description: Hand-grip strength will measure with a J-Tech Medical/USA Tracker Freedom Grip in kg.
Time Frame: as for outcome 1
Population: 12 Wheelchair basketball players and 12 ambulant basketball players Hand Grip test results in baseline, 8 Weeks and 12 Weeks were compared.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Wheelchair Basketball and Ambulant Basketball Players
Number analyzed (Participants) | 24
kg
  Hand Grip Wheelchair Basketball Right Baseline: number analyzed (Participants) | 12
  Hand Grip Wheelchair Basketball Right Baseline | 52.3 (17.5)
  Hand Grip Ambulant Basketball Right Baseline: number analyzed (Participants) | 12
  Hand Grip Ambulant Basketball Right Baseline | 61.6 (11.5)
  Hand Grip Wheelchair Basketball Right 8 Week: number analyzed (Participants) | 12
  Hand Grip Wheelchair Basketball Right 8 Week | 55.6 (16.6)
  Hand Grip Ambulant Basketball Right 8 Week: number analyzed (Participants) | 12
  Hand Grip Ambulant Basketball Right 8 Week | 67.7 (13)
  Hand Grip Wheelchair Basketball Right 12 Week: number analyzed (Participants) | 12
  Hand Grip Wheelchair Basketball Right 12 Week | 53 (16.4)
  Hand Grip Ambulant Basketball Right 12 Week: number analyzed (Participants) | 12
  Hand Grip Ambulant Basketball Right 12 Week | 62.9 (12.4)
  Hand Grip Wheelchair Basketball LeftBaseline: number analyzed (Participants) | 12
  Hand Grip Wheelchair Basketball LeftBaseline | 49.9 (13.7)
  Hand Grip Ambulant Basketball Left Baseline: number analyzed (Participants) | 12
  Hand Grip Ambulant Basketball Left Baseline | 51.9 (11.6)
  Hand Grip Wheelchair Basketball Left 8 Week: number analyzed (Participants) | 12
  Hand Grip Wheelchair Basketball Left 8 Week | 54.6 (13.2)
  Hand Grip Ambulant Basketball Left 8 Week: number analyzed (Participants) | 12
  Hand Grip Ambulant Basketball Left 8 Week | 57.8 (14.9)
  Hand Grip Wheelchair Basketball Left 12 Week: number analyzed (Participants) | 12
  Hand Grip Wheelchair Basketball Left 12 Week | 51.3 (12.9)
  Hand Grip Ambulant Basketball Left 12 Week: number analyzed (Participants) | 12
  Hand Grip Ambulant Basketball Left 12 Week | 53.9 (11.4)

4. Secondary Outcome: Measurement of Range of Motion (Absolute Values Are Being Reported)
Description: Shoulder flexion, abduction and external rotation (E.R), internal rotation (İ.R) range of movement will measure in degrees by J-Tech Medical/US Tracker Freedom Goniometer.
Time Frame: as for outcome 1
Population: 12 Wheelchair basketball players and 12 ambulant basketball players Range of Motion (ROM) measurement results in baseline, 8 Weeks and 12 Weeks were compared.
Measure: Mean (Standard Deviation); unit: Degree
Groups:
- Wheelchair Basketball and Ambulant Basketball Players: 13 players from the North Cyprus Turkcell Wheelchair Basketball Team and 15 players from the Koop Bank Basketball Men's Team voluntarily participated in the study. During evaluations and training, 1 wheelchair basketball player, and 3 stand-up basketball players were excluded from the study as they failed to meet the inclusion criteria. The final participants were 12 male wheelchair basketball players and 12 male stand-up basketball players. After preliminary evaluation, all participants took part in the Throwers Ten exercise programme 3 days a week for 8 weeks. Evaluations were made before the exercise programme, at week 8 at programme completion, and at week 12 after programme completion.
Arm/Group | Wheelchair Basketball and Ambulant Basketball Players
Number analyzed (Participants) | 24
Degree
  ShoulderFlexionWheelchairBasketballRight Baseline: number analyzed (Participants) | 12
  ShoulderFlexionWheelchairBasketballRight Baseline | 161.8 (11.5)
  Shoulder Flexion Ambulant BasketballRight Baseline: number analyzed (Participants) | 12
  Shoulder Flexion Ambulant BasketballRight Baseline | 158.7 (5.5)
  Shoulder Flexion Wheelchair Basketball Right 8Week: number analyzed (Participants) | 12
  Shoulder Flexion Wheelchair Basketball Right 8Week | 159.6 (11.6)
  Shoulder Flexion Ambulant Basketball Right 8Week: number analyzed (Participants) | 12
  Shoulder Flexion Ambulant Basketball Right 8Week | 164.7 (5.8)
  Shoulder Flexion Wheelchair Basketball Right12Week: number analyzed (Participants) | 12
  Shoulder Flexion Wheelchair Basketball Right12Week | 159.3 (11.5)
  Shoulder Flexion Ambulant Basketball Right 12Week: number analyzed (Participants) | 12
  Shoulder Flexion Ambulant Basketball Right 12Week | 161.3 (6)
  ShoulderFlexionWheelchairBasketball Left Baseline: number analyzed (Participants) | 12
  ShoulderFlexionWheelchairBasketball Left Baseline | 158.9 (10.9)
  Shoulder Flexion Ambulant Basketball Left Baseline: number analyzed (Participants) | 12
  Shoulder Flexion Ambulant Basketball Left Baseline | 163.3 (4.8)
  Shoulder Flexion Wheelchair Basketball Left 8 Week: number analyzed (Participants) | 12
  Shoulder Flexion Wheelchair Basketball Left 8 Week | 160.9 (7.5)
  Shoulder Flexion Ambulant Basketball Left 8 Week | 164.4 (6.5)
  Shoulder Flexion Wheelchair Basketball Left 12Week: number analyzed (Participants) | 12
  Shoulder Flexion Wheelchair Basketball Left 12Week | 160.9 (7.5)
  Shoulder Flexion Ambulant Basketball Left 12 Week: number analyzed (Participants) | 12
  Shoulder Flexion Ambulant Basketball Left 12 Week | 165.1 (4.7)
  ShoulderAbductionWheelchairBasketballRightBaseline: number analyzed (Participants) | 12
  ShoulderAbductionWheelchairBasketballRightBaseline | 160.1 (18.1)
  ShoulderAbduction AmbulantBasketballRight Baseline: number analyzed (Participants) | 12
  ShoulderAbduction AmbulantBasketballRight Baseline | 161.6 (7.1)
  ShoulderAbductionWheelchair Basketball Right 8Week: number analyzed (Participants) | 12
  ShoulderAbductionWheelchair Basketball Right 8Week | 162.6 (4.4)
  ShoulderAbduction Ambulant Basketball Right 8Week: number analyzed (Participants) | 12
  ShoulderAbduction Ambulant Basketball Right 8Week | 161.8 (8.5)
  ShoulderAbductionWheelchair Basketball Right12Week: number analyzed (Participants) | 12
  ShoulderAbductionWheelchair Basketball Right12Week | 160.1 (18.3)
  ShoulderAbduction Ambulant Basketball Right 12Week: number analyzed (Participants) | 12
  ShoulderAbduction Ambulant Basketball Right 12Week | 162.8 (9.7)
  ShoulderAbductionWheelchairBasketballLeft Baseline: number analyzed (Participants) | 12
  ShoulderAbductionWheelchairBasketballLeft Baseline | 157.3 (17.8)
  ShoulderAbduction Ambulant BasketballLeft Baseline: number analyzed (Participants) | 12
  ShoulderAbduction Ambulant BasketballLeft Baseline | 162.3 (4.7)
  ShoulderAbductionWheelchair Basketball Left 8Week: number analyzed (Participants) | 12
  ShoulderAbductionWheelchair Basketball Left 8Week | 161.6 (6.2)
  ShoulderAbduction Ambulant Basketball Left 8Week: number analyzed (Participants) | 12
  ShoulderAbduction Ambulant Basketball Left 8Week | 162.7 (5.6)
  ShoulderAbductionWheelchair Basketball Left 12Week: number analyzed (Participants) | 12
  ShoulderAbductionWheelchair Basketball Left 12Week | 157.5 (16.5)
  ShoulderAbduction Ambulant Basketball Left 12Week: number analyzed (Participants) | 12
  ShoulderAbduction Ambulant Basketball Left 12Week | 163.3 (4.6)
  Shoulder E.R Wheelchair Basketball Right Baseline: number analyzed (Participants) | 12
  Shoulder E.R Wheelchair Basketball Right Baseline | 81.7 (10.8)
  Shoulder E.R Ambulant Basketball Right Baseline: number analyzed (Participants) | 12
  Shoulder E.R Ambulant Basketball Right Baseline | 88.8 (12)
  Shoulder E.R Wheelchair Basketball Right 8 Week: number analyzed (Participants) | 12
  Shoulder E.R Wheelchair Basketball Right 8 Week | 85.8 (10.1)
  Shoulder E.R Ambulant Basketball Right 8 Week: number analyzed (Participants) | 12
  Shoulder E.R Ambulant Basketball Right 8 Week | 91.1 (16.3)
  Shoulder E.R Wheelchair Basketball Right 12 Week: number analyzed (Participants) | 12
  Shoulder E.R Wheelchair Basketball Right 12 Week | 81.8 (10.2)
  Shoulder E.R Ambulant Basketball Right 12 Week: number analyzed (Participants) | 12
  Shoulder E.R Ambulant Basketball Right 12 Week | 92.3 (12.5)
  Shoulder E.R Wheelchair Basketball Left Baseline: number analyzed (Participants) | 12
  Shoulder E.R Wheelchair Basketball Left Baseline | 81.7 (10.8)
  Shoulder E.R Ambulant Basketball Left Baseline: number analyzed (Participants) | 12
  Shoulder E.R Ambulant Basketball Left Baseline | 91.2 (9.4)
  Shoulder E.R Wheelchair Basketball Left 8 Week: number analyzed (Participants) | 12
  Shoulder E.R Wheelchair Basketball Left 8 Week | 84.5 (9.4)
  Shoulder E.R Ambulant Basketball Left 8 Week: number analyzed (Participants) | 12
  Shoulder E.R Ambulant Basketball Left 8 Week | 95.3 (8.4)
  Shoulder E.R Wheelchair Basketball Left 12 Week: number analyzed (Participants) | 12
  Shoulder E.R Wheelchair Basketball Left 12 Week | 79.3 (9.7)
  Shoulder E.R Ambulant Basketball Left 12 Week: number analyzed (Participants) | 12
  Shoulder E.R Ambulant Basketball Left 12 Week | 92.4 (9.9)
  Shoulder İ.R Wheelchair Basketball Right Baseline: number analyzed (Participants) | 12
  Shoulder İ.R Wheelchair Basketball Right Baseline | 62.5 (18.6)
  Shoulder İ.R Ambulant Basketball Right Baseline: number analyzed (Participants) | 12
  Shoulder İ.R Ambulant Basketball Right Baseline | 64.8 (8.5)
  Shoulder İ.R Wheelchair Basketball Right 8 Week: number analyzed (Participants) | 12
  Shoulder İ.R Wheelchair Basketball Right 8 Week | 64.1 (13.2)
  Shoulder İ.R Ambulant Basketball Right 8 Week: number analyzed (Participants) | 12
  Shoulder İ.R Ambulant Basketball Right 8 Week | 67.2 (7.6)
  Shoulder İ.R Wheelchair Basketball Right 12 Week: number analyzed (Participants) | 12
  Shoulder İ.R Wheelchair Basketball Right 12 Week | 63.3 (17.4)
  Shoulder İ.R Ambulant Basketball Right 12 Week: number analyzed (Participants) | 12
  Shoulder İ.R Ambulant Basketball Right 12 Week | 65 (8.4)
  Shoulder İ.R Wheelchair Basketball Left Baseline: number analyzed (Participants) | 12
  Shoulder İ.R Wheelchair Basketball Left Baseline | 60.4 (20.1)
  Shoulder İ.R Ambulant Basketball Left Baseline: number analyzed (Participants) | 12
  Shoulder İ.R Ambulant Basketball Left Baseline | 61.8 (11.1)
  Shoulder İ.R Wheelchair Basketball Left 8 Week: number analyzed (Participants) | 12
  Shoulder İ.R Wheelchair Basketball Left 8 Week | 66.9 (14.6)
  Shoulder İ.R Ambulant Basketball Left 8 Week: number analyzed (Participants) | 12
  Shoulder İ.R Ambulant Basketball Left 8 Week | 71.2 (10.9)
  Shoulder İ.R Wheelchair Basketball Left 12 Week: number analyzed (Participants) | 12
  Shoulder İ.R Wheelchair Basketball Left 12 Week | 63.3 (17.4)
  Shoulder İ.R Ambulant Basketball Left 12 Week: number analyzed (Participants) | 12
  Shoulder İ.R Ambulant Basketball Left 12 Week | 63 (11.7)

ADVERSE EVENTS:
Time Frame: Measurements data were collected at the begining of the study, 8 Weeks of the study and 12 Weeks of the study.
Description: Not including serious adverse events. 4 participants were affected from musculoskeletal pain (other adverse event) and they were excluded from the study. Protocol enrollment was 28, because of excluding 4 participants, participant flow number was 24.
Groups:
- Wheelchair Basketball and Ambulant Basketball Players: 13 players from the North Cyprus Turkcell WC Basketball Team and 15 players from the Koop Bank Basketball Men's Team voluntarily participated in the study. During evaluations and training, one WC basketball player, and three stand-up basketball players were excluded from the study as they failed to meet the inclusion criteria. The final participants were 12 male WC basketball players and 12 male stand-up basketball players. After preliminary evaluation, all participants took part in the Throwers Ten exercise programme 3 days a week for 8 weeks. Evaluations were made before the exercise programme, at week 8 in programme completion, and at week 12 after programme completion.
Arm/Group | Wheelchair Basketball and Ambulant Basketball Players
All-Cause Mortality (participants affected / at risk) | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 4/28
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Wheelchair Basketball and Ambulant Basketball Players (N=28)
Pain (Musculoskeletal and connective tissue disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-20): https://cdn.clinicaltrials.gov/large-docs/90/NCT04019990/Prot_SAP_000.pdf